CLINICAL TRIAL: NCT01533961
Title: Randomized, Double-blind, Placebo-controlled Sequential Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SCYX-7158 After Single Oral Ascending Doses in Healthy Male Volunteers
Brief Title: Human African Trypanosomiasis: First in Man Clinical Trial of a New Medicinal Product, the SCYX-7158
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNDiOXA001; 2011-004639-30 (EudraCT Number)
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2012-02

CONDITIONS: Trypanosomiasis; Trypanosomiasis, African; Protozoan Infections; Parasitic Diseases
Keywords: neglected disease; africa; new drug; oral drug; parasite
MeSH Terms: conditions — Trypanosomiasis; Trypanosomiasis, African; Protozoan Infections; Parasitic Diseases; Neglected Diseases | interventions — SCYX 7158

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCYX-7158 (Experimental): In each dose group (8 subjects) , 6 Healthy Volunteers receive SCYX-7158
  Interventions: Drug: SCYX-7158
- Placebo of SCYX-7158 (Placebo Comparator): In each dose group (8 subjects) , 2 Healthy Volunteers receive placebo of SCYX-7158
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCYX-7158
  Arms: SCYX-7158
Drug: Placebo
  Arms: Placebo of SCYX-7158

SUMMARY:
This study is aimed at assessing the tolerability and pharmacokinetic parameters of SCYX-7158 in healthy volunteers. In animal models of both acute and chronic experimental Trypanosomiasis infections, SCYX-7158 shows highly promising efficacy.

DETAILED DESCRIPTION:
The present study is designed to obtain safety, tolerability and PK data after single oral administration of increasing doses of SCYX-7158 in healthy male sub-Saharan African subjects. This study will also assess the impact on the relative bioavailability of SCYX-7158 administered as a capsule after single oral dose administration.

The study will be divided in 3 different parts. Study Part I will be a randomized, double-blind, placebo-controlled, single ascending dose study with SCYX-7158 administered as a capsule.

A other part is scheduled to evaluate the impact of activated charcoal intake on the PK characteristics of SCYX-7158 and determine the most adapted treatment schedule for charcoal to enhance SCYX-7158 elimination while allowing a sustained drug exposure likely to be therapeutically active.

A last part is planned to evaluate the pharmacokinetics of a new formulation (tablet) of SCYX-7158 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteers 18 to 45 years of age,
* All subjects to be of sub-Saharan African origins with both parents of Sub-Saharan African origins too,
* Male subjects with a body mass index (BMI) calculated as weight in kg/(height in m2) from 18 to 28 kg/m2 at screening,
* Able to communicate well with the Investigator and research staff and to comply with the requirements of the entire study,
* Provision of written informed consent to participate as shown by a signature on the volunteer consent form,
* Light smokers (less than 5 cigarettes per day) or subjects who are non-smokers. No smoking (or use of smoking substitute e.g. nicotine patch) is permitted from screening throughout the study,
* Normal arterial blood pressure (BP) and pulse rate or, if abnormal, considered not clinically significant by the principal Investigator. These will be measured after resting for 5 min.
* Registered with the French Social Security in agreement with the French law on biomedical experimentation.

Exclusion Criteria:

* Who on direct questioning and physical examination have evidence of any clinically significant acute or chronic disease, including known or suspected HIV, HBV or HCV infection,
* Who previously received SCYX-7158,
* Who presented acute or chronic or history of symptoms of Gastro intestinal disturbances (GI) or on physical examination have evidence of any clinical signs of acute or chronic GI abnormality ( i.e hemorrhoids, GI bleeding…)
* With any clinically significant abnormality following review of pre-study laboratory tests (aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) must be within normal ranges), vital signs, full physical examination and ECG,
* Who are within the exclusion period defined in the National Register for Healthy Volunteers of the French Ministry of Health,
* Who forfeit their freedom by administrative or legal award or who were under guardianship,
* Unwilling to give their informed consent,
* Who have a positive laboratory test for Hepatitis B surface antigen (HbsAg), or anti-HIV 1/2 or anti- HCV antibodies
* Who have a history of allergy, intolerance or photosensitivity to any drug,
* Who have a history of serious allergy, asthma, allergic skin rash or sensitivity to any drug,
* Who are known or suspected alcohol or drug abusers (more than 14 units of alcohol per week, one unit = 8 g or about 10 mL of pure alcohol),
* Who drink more than 8 cups daily of beverage containing caffeine,
* Who have a positive laboratory test for urine drug screening (opiates, cocaine, amphetamine, cannabis, benzodiazepines),
* Who have undergone surgery or have donated blood within 12 weeks prior to the start of the study,
* Who have taken any prescribed or over the counter drug (including antacid drug), with the exception of paracetamol (up to 3 g per day) within 2 weeks prior to the first dose administration,
* Who have any clinical condition or prior therapy which, in the opinion of the Investigator, made the subject unsuitable for the study,
* Who participated to any clinical trial with an investigational drug in the past 3 months preceding study entry.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2012-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Occurence of adverse events (AEs) | 9 to 37 days, depending on the part of the study
  Monitoring for the occurrence of AEs. Changes in physical examination, vital signs (blood pressure and pulse rate), ECG, and clinical laboratory tests (biochemistry, hematology, and urinalysis).

SECONDARY OUTCOMES:
Pharmacokinetic (blood concentration of SCYX-7158 and metabolite) | from pre-dose until 168 h post-dose.
Pharmacokinetic (urine concentration of SCYX-7158 and metabolite) | from pre-dose until 168 h post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Tarral, MD, Study Director — Drugs for Neglected Diseases initiative
Locations (2):
- France (2):
  - Optimed, Grenoble
  - SGS Aster, Paris

REFERENCES:
- [Derived] Tarral A, Hovsepian L, Duvauchelle T, Donazzolo Y, Latreille M, Felices M, Gualano V, Delhomme S, Valverde Mordt O, Blesson S, Voiriot P, Strub-Wourgaft N. Determination of the Optimal Single Dose Treatment for Acoziborole, a Novel Drug for the Treatment of Human African Trypanosomiasis: First-in-Human Study. Clin Pharmacokinet. 2023 Mar;62(3):481-491. doi: 10.1007/s40262-023-01216-8. Epub 2023 Feb 10. PMID 36763327
- See also: Sponsor website — http://www.dndi.org